CLINICAL TRIAL: NCT06173258
Title: Evaluation of Artificial Intelligence for Adenoma Detection in Water Exchange Colonoscopy: the WEAID Randomized Controlled Trial (Water Exchange With Artificial Intelligence-assisted Detection)
Brief Title: Water Exchange Colonoscopy With Artificial Intelligence-assisted Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evergreen General Hospital, Taiwan (Other)
Collaborators: Digestive Endoscopy Unit, CTO Hospital, Iglesias, Italy (Unknown); The Sepulveda Ambulatory Care Center, VAGLAHS, UCLA in the USA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: WEAID
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Colon Adenoma; Colonoscopy; Colon Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water exchange alone (Active Comparator): Residual air in the colon will be removed, water will be infused to guide insertion through an airless lumen. Infused water will be removed by suction, along with residual fecal debris, predominantly during insertion.
  Interventions: Device: Water exchange alone; Device: Water exchange plus Artificial Intelligence (AI)
- Water exchange plus Artificial intelligence (AI) (Experimental): During colonoscopic insertion, residual air in the colon will be removed, water will be infused to guide insertion through an airless lumen. Infused water will be removed by suction, along with residual fecal debris, predominantly during insertion. A commercially available AI system (CAD-EYE, Fujifilm, used in Taiwan; Endo-AID, Olympus used in Italy) will be employed. During AI-assisted procedures, the AI will be activated during the withdrawal phase of the procedure, providing a bounding box as output any time a lesion that is suspected to be a polyp is recognized by the AI device.
  Interventions: Device: Water exchange alone; Device: Water exchange plus Artificial Intelligence (AI)

INTERVENTIONS:
Device: Water exchange alone — During the insertion phase of water exchange colonoscopy, the air pump will be turned off, while the colon will be irrigated with warm-to-touch water using a flushing pump. The water exchange approach involves the simultaneous infusion of water to facilitate luminal expansion and suction of unclean water during insertion. Upon reaching the cecum, where most of the water is suctioned to collapse the cecal lumen, the air pump will be opened. Withdrawal from the cecum will begin in the left lateral position. Similar withdrawal techniques with adequate luminal distention and comprehensive examination behind the folds will be emphasized. Any position change away from the original left lateral position in any colon segment during the withdrawal phase will be recorded. Tandem examination of specific colon segments, including the right colon, either in the standard modality or retroflexion, is prohibited.
Device: Water exchange plus Artificial Intelligence (AI) — Similar water exchange technique as the active comparator will be employed during insertion. Similar withdrawal inspection techniques as the active comparator will be used. During withdrawal phase, commercially available AI system (CAD-EYE, Fujifilm, EU and Taiwan; Endo-AID, Olympus, EU and Taiwan) will be activated, providing a bounding box as output any time a lesion that is suspected to be a polyp is recognized by the AI device. False positive activation is defined as the identification by AI systems of an area during the withdrawal phase that is not deemed to be a colorectal lesion after re-examination by the colonoscopist. Real-time flagging of FP activation will be recorded by investigators and study staff.

SUMMARY:
The goal of this clinical trial is to compare the detected adenoma per colonoscopy (APC) in participants undergoing screening, surveillance, and positive fecal immunochemical test (FIT) or guaiac fecal occult blood test (gFOBT). There will be two arms in this study: WE water control and water plus artificial intelligence (AI). The main question it aims to answer is whether the addition of AI into water exchange (WE) colonoscopy increases APC than WE alone. The control method will use water instead of air inserted into the colon. The study method will use a commercially available AI system plus water during the procedure. Researchers will compare APCs to see if the addition of AI increases detection of adenomas during WE colonoscopy.

DETAILED DESCRIPTION:
This will be a multi-site, multi-national, unblinded investigators, prospective Random Control Trial (RCT). Randomization (1:1 to WE alone and WE-AI) will be based on computer generated random numbers placed inside opaque sealed envelopes. The envelope (in pre-arranged order) will be opened to reveal the code when the colonoscopist is ready to insert the endoscope to begin the examination. This will be a comparison of two different methods with two arms (WE, WE-AI) to see which one is better at detecting adenomas.

Patient recruitment will be conducted at three hospitals in Italy and Taiwan: Digestive Endoscopy Unit, CTO Hospital, Iglesias, Italy; Digestive Endoscopy and Gastroenterology Unit, Manzoni Hospital, Lecco, Italy; Evergreen General Hospital, Taoyuan, Taiwan. The Sepulveda Ambulatory Care Center, VAGLAHS, UCLA in the USA will be a non-recruiting participating site. The study period is expected to be 3 years (from November 2023 to October 2026).

Patients aged 45-75 y/o at average risk of colorectal cancer who are willing to participate will sign an informed consent before starting the colonoscopy procedure. Separate parallel randomization will be set up at each site, stratified by investigator and type of colonoscopy (primary screening, surveillance, or positive FIT or gFOBT). Mode of sedation will include unsedated, on demand sedation, conscious sedation or full sedation with propofol. Randomization will be carried out by computer-generated sequences using a block design (four participants per block).

Control Method: One arm of the study will include sedated/unsedated colonoscopy with water (WE) as the control method. Residual air in the colon will be removed and water will be infused to guide insertion through an airless lumen. Infused water will be removed by suction, along with residual fecal debris, predominantly during insertion.

Study method: The other arm entail the addition of a commercially available AI system (CAD-EYE, Fujifilm; Endo-AID, Olympus) to the high-definition colonoscopy system. This arm includes sedated/unsedated colonoscopy with AI detection device plus water (WE).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 45-75 years at average risk for colorectal cancer who plan to undergo colonoscopy for primary screening, postpolypectomy surveillance, and individuals with positive fecal immunochemical test or guaiac fecal occult blood test results.

Exclusion Criteria:

* Patients with a history of inflammatory bowel disease
* Patients with hereditary colorectal cancer syndrome or serrated polyposis syndrome
* Patients with a personal history of colorectal cancer
* Patients with a history of colorectal resection
* Patients with colonic stricture
* Patient with severe comorbid illnesses rendering polypectomy unsafe
* Patients with colonoscopy contraindications (e.g., acute diverticulitis or toxic megacolon)
* Therapeutic colonoscopy (e.g., hemostasis, removal of a large polyp)
* Emergent colonoscopy
* Pregnant women or those planning pregnancy
* Patients unwilling to participate in the study

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
Adenoma per colonoscopy | One week (after the colonoscopy procedure, when pathology report is released)
  Adenoma per colonoscopy is calculated as the total number of adenomas detected divided by the total number of colonoscopies performed in the subjects undergoing a complete colonoscopy.
Adenoma detection rate | One week (after the colonoscopy procedure, when pathology report is released)
  The percentage of subjects undergoing a complete colonoscopy, who have at least one histologically confirmed adenoma detected and removed.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Cadoni, MD, Principal Investigator — Endoscopy Digestive Unit, CTO Hospital, Iglesias, Italy
Locations (2):
- CTO Hospital, Iglesias, Italy
- Chi-Liang Cheng, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wieszczy P, Bugajski M, Januszewicz W, Rupinska M, Szlak J, Pisera M, Turkot MH, Rupinski M, Wojciechowska U, Didkowska J, Regula J, Kaminski MF. Comparison of Quality Measures for Detection of Neoplasia at Screening Colonoscopy. Clin Gastroenterol Hepatol. 2023 Jan;21(1):200-209.e6. doi: 10.1016/j.cgh.2022.03.023. Epub 2022 Mar 24. PMID 35341951
- [Background] Denis B, Sauleau EA, Gendre I, Piette C, Bretagne JF, Perrin P. Measurement of adenoma detection and discrimination during colonoscopy in routine practice: an exploratory study. Gastrointest Endosc. 2011 Dec;74(6):1325-36. doi: 10.1016/j.gie.2011.07.038. Epub 2011 Sep 29. PMID 21958899
- [Background] Cadoni S, Falt P, Rondonotti E, Radaelli F, Fojtik P, Gallittu P, Liggi M, Amato A, Paggi S, Smajstrla V, Urban O, Erriu M, Koo M, Leung FW. Water exchange for screening colonoscopy increases adenoma detection rate: a multicenter, double-blinded, randomized controlled trial. Endoscopy. 2017 May;49(5):456-467. doi: 10.1055/s-0043-101229. Epub 2017 Mar 10. PMID 28282689
- [Background] Hsieh YH, Tseng CW, Hu CT, Koo M, Leung FW. Prospective multicenter randomized controlled trial comparing adenoma detection rate in colonoscopy using water exchange, water immersion, and air insufflation. Gastrointest Endosc. 2017 Jul;86(1):192-201. doi: 10.1016/j.gie.2016.12.005. Epub 2016 Dec 15. PMID 27988288
- [Background] Hassan C, Spadaccini M, Mori Y, Foroutan F, Facciorusso A, Gkolfakis P, Tziatzios G, Triantafyllou K, Antonelli G, Khalaf K, Rizkala T, Vandvik PO, Fugazza A, Rondonotti E, Glissen-Brown JR, Kamba S, Maida M, Correale L, Bhandari P, Jover R, Sharma P, Rex DK, Repici A. Real-Time Computer-Aided Detection of Colorectal Neoplasia During Colonoscopy : A Systematic Review and Meta-analysis. Ann Intern Med. 2023 Sep;176(9):1209-1220. doi: 10.7326/M22-3678. Epub 2023 Aug 29. PMID 37639719
- [Background] Mori Y, Wang P, Loberg M, Misawa M, Repici A, Spadaccini M, Correale L, Antonelli G, Yu H, Gong D, Ishiyama M, Kudo SE, Kamba S, Sumiyama K, Saito Y, Nishino H, Liu P, Glissen Brown JR, Mansour NM, Gross SA, Kalager M, Bretthauer M, Rex DK, Sharma P, Berzin TM, Hassan C. Impact of Artificial Intelligence on Colonoscopy Surveillance After Polyp Removal: A Pooled Analysis of Randomized Trials. Clin Gastroenterol Hepatol. 2023 Apr;21(4):949-959.e2. doi: 10.1016/j.cgh.2022.08.022. Epub 2022 Aug 28. PMID 36038128
- [Background] Nehme F, Coronel E, Barringer DA, Romero LG, Shafi MA, Ross WA, Ge PS. Performance and attitudes toward real-time computer-aided polyp detection during colonoscopy in a large tertiary referral center in the United States. Gastrointest Endosc. 2023 Jul;98(1):100-109.e6. doi: 10.1016/j.gie.2023.02.016. Epub 2023 Feb 18. PMID 36801459
- [Background] Tang CP, Lin TL, Hsieh YH, Hsieh CH, Tseng CW, Leung FW. Polyp detection and false-positive rates by computer-aided analysis of withdrawal-phase videos of colonoscopy of the right-sided colon segment in a randomized controlled trial comparing water exchange and air insufflation. Gastrointest Endosc. 2022 Jun;95(6):1198-1206.e6. doi: 10.1016/j.gie.2021.12.020. Epub 2021 Dec 30. PMID 34973967
- [Background] Patel SG, May FP, Anderson JC, Burke CA, Dominitz JA, Gross SA, Jacobson BC, Shaukat A, Robertson DJ. Updates on Age to Start and Stop Colorectal Cancer Screening: Recommendations From the U.S. Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2022 Jan;162(1):285-299. doi: 10.1053/j.gastro.2021.10.007. Epub 2021 Nov 15. PMID 34794816
- [Background] Saftoiu A, Hassan C, Areia M, Bhutani MS, Bisschops R, Bories E, Cazacu IM, Dekker E, Deprez PH, Pereira SP, Senore C, Capocaccia R, Antonelli G, van Hooft J, Messmann H, Siersema PD, Dinis-Ribeiro M, Ponchon T. Role of gastrointestinal endoscopy in the screening of digestive tract cancers in Europe: European Society of Gastrointestinal Endoscopy (ESGE) Position Statement. Endoscopy. 2020 Apr;52(4):293-304. doi: 10.1055/a-1104-5245. Epub 2020 Feb 12. PMID 32052404
- [Background] Rex DK, Schoenfeld PS, Cohen J, Pike IM, Adler DG, Fennerty MB, Lieb JG 2nd, Park WG, Rizk MK, Sawhney MS, Shaheen NJ, Wani S, Weinberg DS. Quality indicators for colonoscopy. Gastrointest Endosc. 2015 Jan;81(1):31-53. doi: 10.1016/j.gie.2014.07.058. Epub 2014 Dec 2. No abstract available. PMID 25480100
- [Background] Kaminski MF, Thomas-Gibson S, Bugajski M, Bretthauer M, Rees CJ, Dekker E, Hoff G, Jover R, Suchanek S, Ferlitsch M, Anderson J, Roesch T, Hultcranz R, Racz I, Kuipers EJ, Garborg K, East JE, Rupinski M, Seip B, Bennett C, Senore C, Minozzi S, Bisschops R, Domagk D, Valori R, Spada C, Hassan C, Dinis-Ribeiro M, Rutter MD. Performance measures for lower gastrointestinal endoscopy: a European Society of Gastrointestinal Endoscopy (ESGE) quality improvement initiative. United European Gastroenterol J. 2017 Apr;5(3):309-334. doi: 10.1177/2050640617700014. Epub 2017 Mar 16. PMID 28507745
- [Background] Kaltenbach T, Gawron A, Meyer CS, Gupta S, Shergill A, Dominitz JA, Soetikno RM, Nguyen-Vu T, A Whooley M, Kahi CJ. Adenoma Detection Rate (ADR) Irrespective of Indication Is Comparable to Screening ADR: Implications for Quality Monitoring. Clin Gastroenterol Hepatol. 2021 Sep;19(9):1883-1889.e1. doi: 10.1016/j.cgh.2021.02.028. Epub 2021 Feb 19. PMID 33618027
- [Background] Hassan C, East J, Radaelli F, Spada C, Benamouzig R, Bisschops R, Bretthauer M, Dekker E, Dinis-Ribeiro M, Ferlitsch M, Fuccio L, Awadie H, Gralnek I, Jover R, Kaminski MF, Pellise M, Triantafyllou K, Vanella G, Mangas-Sanjuan C, Frazzoni L, Van Hooft JE, Dumonceau JM. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2019. Endoscopy. 2019 Aug;51(8):775-794. doi: 10.1055/a-0959-0505. Epub 2019 Jul 11. PMID 31295746
- [Background] Hassan C, Badalamenti M, Maselli R, Correale L, Iannone A, Radaelli F, Rondonotti E, Ferrara E, Spadaccini M, Alkandari A, Fugazza A, Anderloni A, Galtieri PA, Pellegatta G, Carrara S, Di Leo M, Craviotto V, Lamonaca L, Lorenzetti R, Andrealli A, Antonelli G, Wallace M, Sharma P, Rosch T, Repici A. Computer-aided detection-assisted colonoscopy: classification and relevance of false positives. Gastrointest Endosc. 2020 Oct;92(4):900-904.e4. doi: 10.1016/j.gie.2020.06.021. Epub 2020 Jun 16. PMID 32561410
- [Background] Spadaccini M, Hassan C, Alfarone L, Da Rio L, Maselli R, Carrara S, Galtieri PA, Pellegatta G, Fugazza A, Koleth G, Emmanuel J, Anderloni A, Mori Y, Wallace MB, Sharma P, Repici A. Comparing the number and relevance of false activations between 2 artificial intelligence computer-aided detection systems: the NOISE study. Gastrointest Endosc. 2022 May;95(5):975-981.e1. doi: 10.1016/j.gie.2021.12.031. Epub 2022 Jan 4. PMID 34995639

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT06173258/Prot_SAP_000.pdf